CLINICAL TRIAL: NCT06705660
Title: Investigation of the Effects of WEB-based Lifestyle Training and Progressive Relaxation Training in Women With Premenstrual Syndrome: 4-Week Follow-up Randomized Controlled Trial
Brief Title: Effect of Web-Based Life Style Training and Relaxation Training in Women With Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysenur KARAKUS (Other)
Responsible Party: Sponsor-Investigator, Aysenur KARAKUS, Lecturer, Çankırı Karatekin University
Organization: Çankırı Karatekin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PMSWWEB
Record Dates: First submitted 2024-10-09; First posted 2024-11-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome; Lifestyle; Relaxation; Women
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: Within the scope of the study, women with Premenstrual Syndrome (PMS) will be divided into three groups. The first group will receive web-based lifestyle interventions, while the second group will be given web-based progressive relaxation training. The third group will serve as the control group and will not receive any training. Assessments will be planned at two stages: before the intervention (baseline assessments) and after the intervention (8 weeks later). The web-based lifestyle interventions and progressive relaxation training will be provided by monitoring the participants' menstrual cycles, ensuring that the training is administered over two menstrual cycles. Evaluations will be conducted both before and after the training periods, and an additional follow-up assessment will be performed one month (4 weeks later-the next cycle) after the completion of the training, to monitor the effects. This approach aims to observe the long-term outcomes of the training.
Who Masked: Outcomes Assessor
Masking Description: Statistician blinding method will be applied to perform statistical analyses objectively. In this way, the statistician will not know which participant belongs to which group, thereby increasing the objectivity and reliability of the analysis results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- WEB-based lifestyle interventions (Active Comparator): The web-based lifestyle interventions will be administered to women by monitoring their menstrual cycles for 8 weeks, with sessions held twice a week for 30-45 minutes each (totaling 16 sessions). Measurements will be taken both before the intervention and after its completion. An additional measurement will be conducted during the following menstrual cycle, 4 weeks later, to ensure follow-up.In this study, telehealth and counseling services will be provided. Through telehealth and counseling, women will have the opportunity to communicate online with healthcare professionals and receive guidance on health goals, nutrition, exercise, and stress management
  Interventions: Other: The WEB-based lifestyle interventions
- Control Group (No Intervention): The third group will serve as the control group and will not receive any training.
- The WEB-based progressive relaxation training (Active Comparator): WEB-based progressive relaxation training will be given for 8 weeks, 2 days a week for 30-45 minutes (16 sessions), following the menstrual cycles of women. Measurements will be taken before and after (at the end of) the intervention. Measurements will be taken 4 weeks after the next menstrual cycle to ensure follow-up.
  Progressive relaxation training is an easy-to-learn, non-invasive and side-effect free method. PGE beginners will be trained for at least 30 minutes and practitioners who have learned the basics of the method will be trained to introduce PGE for 15 minutes. Prior to the PGE, individuals will be informed that they should not come overly hungry or overly full (eating should be finished 2 hours before), wear loose and comfortable clothes, avoid clothes that tightly wrap the abdomen (pants, dresses, belts), remove contact lenses, glasses, jewelry and tight shoes. PGE will be administered in a quiet, comfortable and dimly lit place. Women will perform PCI in the supine posi
  Interventions: Other: WEB-based progressive relaxation training

INTERVENTIONS:
Other: WEB-based progressive relaxation training — WEB-based progressive relaxation training will be given for 8 weeks, 2 days a week for 30-45 minutes (16 sessions), following the menstrual cycles of women. Measurements will be taken before and after (at the end of) the intervention. Measurements will be taken 4 weeks after the next menstrual cycle to ensure follow-up.
  Progressive relaxation training is an easy-to-learn, non-invasive and side-effect free method. PGE beginners will be trained for at least 30 minutes and practitioners who have learned the basics of the method will be trained to introduce PGE for 15 minutes. Prior to the PGE, individuals will be informed that they should not come overly hungry or overly full (eating should be finished 2 hours before), wear loose and comfortable clothes, avoid clothes that tightly wrap the abdomen (pants, dresses, belts), remove contact lenses, glasses, jewelry and tight shoes. PGE will be administered in a quiet, comfortable and dimly lit place. Women will perform PCI in the supine posit
  Arms: The WEB-based progressive relaxation training
Other: The WEB-based lifestyle interventions — The WEB-based lifestyle interventions will be administered to women by monitoring their menstrual cycles for 8 weeks, with sessions held twice a week for 30-45 minutes each (totaling 16 sessions). Measurements will be taken both before the intervention and after its completion. An additional measurement will be conducted during the following menstrual cycle, 4 weeks later, to ensure follow-up.In this study, telehealth and counseling services will be provided. Through telehealth and counseling, women will have the opportunity to communicate online with healthcare professionals and receive guidance on health goals, nutrition, exercise, and stress management
  Arms: WEB-based lifestyle interventions

SUMMARY:
The aim of this study is to investigate the effectiveness of web-based lifestyle education and progressive relaxation training provided to women with PMS.

During menstruation, an important indicator of reproductive health, women encounter various problems. One of these problems is premenstrual syndrome (PMS). PMS is characterized by its occurrence in 30-40% of women of reproductive age, beginning in the late luteal phase of their menstrual cycle, and presenting with a series of physical, psychological, emotional, behavioral, and social symptoms that end with menstruation. Common symptoms of PMS include changes in appetite, irritability, depression, anxiety, difficulty concentrating, headaches, weight gain, constipation, fatigue, abdominal and lower back pain, breast swelling and tenderness, and mood swings. These symptoms negatively affect the quality of life and participation in social and family activities of women with PMS. Moreover, it leads to reduced productivity in the workforce, lower quality of work life, economic losses, and increased accident potential. Additionally, it has been observed to negatively impact young women's self-esteem, school attendance if they are students, academic success, and willingness to engage in hobbies, thereby affecting their participation in meaningful and purposeful activities-referred to as occupations. Managing lifestyle changes and controlling symptoms in PMS is only possible through behavior change. Recent studies have focused on web-based lifestyle interventions and progressive relaxation training (PRT) to promote behavior change in PMS. The accessibility, ease of use, cost/time efficiency, centralization of user health data, and the ability to update remotely make web-based applications a preferred option in health interventions.

In this study, women with PMS will be divided into three groups. The first group will receive web-based lifestyle interventions, the second group will receive web-based PRT, and the third group will serve as a control group without any education. Web-based lifestyle interventions and PRT will be provided by tracking the menstrual cycles of the women. Both interventions will be delivered over the course of two menstrual cycles. A follow-up assessment will be conducted one month after the completion of the trainings (4 weeks later, during the next cycle). Assessments will be planned for both before the intervention (baseline assessment) and after the intervention (8 weeks later). The women's sociodemographic and clinical characteristics related to menstruation will be assessed with the Sociodemographic and Clinical Information Form, their type and severity of premenstrual symptoms with the Premenstrual Syndrome Scale, their anxiety and stress levels with the Hospital Anxiety and Stress Scale, their quality of life with the Nottingham Health Profile, their occupational performance and participation with the Canadian Occupational Performance Measure, and their occupational satisfaction with the Occupational Balance Questionnaire.

DETAILED DESCRIPTION:
Improving and maintaining health and quality of life in women is possible by protecting reproductive health . Menstruation, an important indicator of reproductive health, is a significant process that continues from adolescence to menopause in women. Women may encounter various problems related to the menstruation process . One of the most important of these problems is premenstrual syndrome (PMS) .

Premenstrual syndrome is seen in 30-40% of women of reproductive age and is characterized by a series of physical, psychological, emotional, behavioral, and social symptoms that begin in the late luteal phase of their menstrual cycle. These symptoms typically begin in the luteal phase and end within a few days after menstruation. Common symptoms of PMS include changes in appetite, irritability, depression, anxiety, difficulty concentrating, headaches, weight gain, constipation, fatigue, abdominal and lower back pain, breast swelling and tenderness, and mood swings. The cyclical nature of symptom changes is one of the syndrome's notable features. Although the etiology of PMS is uncertain, it is thought that the common symptoms may largely result from sex steroids secreted during the luteal phase and the serotonin mechanism in the central nervous system .

PMS causes a decrease in workforce productivity and the quality of work life, leading to economic losses and an increase in accident potential. In addition, these symptoms have been observed to reduce young women's self-esteem, school attendance (if they are students), academic success, and desire to engage in hobbies, thus negatively affecting their participation in meaningful and purposeful activities, also known as occupations . A study by Park et al. (2023) identified three problematic areas in women with PMS: occupational disruption, social disruption, and a decrease in self-awareness while engaging in their occupations. Additionally, it has been observed that PMS symptoms interfere with women's ability to perform their occupations, including self-care, productivity, and leisure, thereby disrupting their routines and interpersonal relationships. Other studies, such as one by Süt et al. (2006), found that PMS decreased work-related quality of life in working women (n=134). In another study by Victor et al. (2019), conducted with female students (n=634) in Brazil, it was found that students with PMS had lower quality of life and academic achievement compared to asymptomatic students. Similarly, a study conducted with female students (n=235) in Northern India found a moderate correlation between PMS and health-related quality of life (Bhuvaneswari et al., 2019). Additionally, it was reported that premenstrual symptoms negatively impacted daily life activities, learning activities, and even communication with friends and family. Thus, creating an effective and widespread intervention protocol for PMS, which imposes a socioeconomic burden and negatively affects occupational participation and quality of life in women, is of great importance.

Occupational therapy is a health profession that promotes lifestyle changes and habits that enhance health, facilitating participation in meaningful and purposeful activities. Non-pharmacological methods aimed at alleviating the physical and psychiatric symptoms of PMS, such as yoga, Pilates, aerobic exercises, electrotherapy, and cognitive-behavioral therapy, have been used. One of the important methods used in PMS management is lifestyle change interventions aimed at instilling and maintaining behaviors such as diet, sleep hygiene, and exercise. A randomized controlled trial conducted by Alyazkaya et al. (2020) demonstrated that lifestyle education based on the health belief model reduced PMS symptoms. Similarly, a randomized controlled trial by Yılmaz & Aydın (2019) found that diet and exercise reduced PMS symptoms. Studies have emphasized the importance of expanding the scope of interventions that include lifestyle changes. Thus, it is important to expand the impact of lifestyle interventions on PMS symptoms and compare them with different interventions.

Controlling lifestyle changes and symptoms in PMS is only possible through behavior change. Recent studies have suggested the use of various tools (mobile-based, tele-rehabilitation, phone) to promote behavior change in PMS. Among these tools, one of the most noteworthy is web-based lifestyle interventions. Web-based applications are preferred in healthcare interventions due to their accessibility, ease of use, cost/time efficiency, centralization of user health data, and the ability to update remotely.However, studies on web-based lifestyle change interventions in women with PMS are limited (Bastani & Hashemi, 2012). In a study by Bastani & Hashemi (2012), web-based lifestyle change education was found to improve general health and well-being in university students with PMS after the intervention. Therefore, further studies are needed to understand and expand the use of web-based lifestyle education in PMS.

Another method for addressing premenstrual syndrome is progressive relaxation training (PRT). Progressive relaxation training involves gradually tensing and relaxing muscle groups in 16 areas of the body. It has been reported that PRT reduces stress, depression, and pain, while improving sleep and quality of life. In a randomized controlled trial conducted by Abic et al. (2024) with women with PMS (n=68), yoga and PRT were provided to manage PMS-related depression, anxiety, and stress. It was found that PRT combined with yoga reduced PMS symptoms. Thirupathi's (2017) study of 60 young adult women revealed that PRT reduced PMS symptoms and improved quality of life. In another study by Rausch et al. (2006) with 387 women, PRT was found to reduce cognitive, somatic, and general anxiety. Studies have highlighted the need for expanding the use of progressive relaxation training within treatment protocols. In this context, studies on the use of PRT for PMS symptoms are gaining importance.

In the literature, web-based PRT applications have been used in various disease populations (caregivers, women with migraines, individuals with back pain, healthcare workers, office workers). However, studies on women with PMS are limited and few. In a study by Marfuah et al. (2021), progressive relaxation training was provided to adolescent women (n=52) through a mobile application, and it was found that PRT reduced PMS symptoms and that more interventions focused on reproductive health were needed for young women.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 years Menstrual cycle length within normal limits (21-35 days) Presence of premenstrual symptoms Willingness to participate in the study

Exclusion Criteria:

* Receiving medical or rehabilitative treatment for PMS within the last 6 months
* Suspected pregnancy or history of childbirth
* Use of an intrauterine device
* History of surgery involving the abdominal, pelvic region, and/or spine within the last year
* Use of surgical contraceptives or antidepressants within the last 6 months
* Presence of a diagnosed severe spinal deformity such as scoliosis or any pathology involving the spine (e.g., disc herniation, spondylolisthesis)
* Presence of neurological (headache or migraine), rheumatological, or mental health conditions
* Existence of a cardiopulmonary disease (e.g., Chronic Obstructive Pulmonary Disease, chronic heart failure)
* Body Mass Index (BMI) ≥ 30 kg/m²
* Undergoing treatment for insomnia
* Presence of a dermatological condition (e.g., allergies, psoriasis)
* Difficulty in communicating in Turkish

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The population of the study consists of women, while the sample will be comprised of women aged 18-35 who have Premenstrual Syndrome (PMS). The study group will be formed from women who agree to participate in the study."
Enrollment: 66 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
The Premenstrual Syndrome Scale (PMSS) | From enrollment to the end of treatment at 8 weeks
  The Premenstrual Syndrome Scale (PMSS) is a 44-item, five-point Likert-type scale (ranging from 'Never' to 'Always') developed to determine the type and severity of PMS symptoms. As stated in the instructions at the beginning of the scale, after reading each item, participants mark their response based on how often they experience that symptom 'within the week before menstruation.' The scoring of the scale assigns points as follows: 'Never' = 1 point, 'Rarely' = 2 points, 'Sometimes' = 3 points, 'Often' = 4 points, and 'Always' = 5 points. The lowest possible score on the scale is 44, and the highest possible score is 220. Based on the scores obtained from the scale, PMS severity can be categorized. A total score of 88 or above indicates severe PMS symptoms, while a score below 88 indicates mild PMS symptoms (Gençdoğan, 2006). In the development study of the scale, Gençdoğan (2006) reported a Cronbach's alpha value of 0.75.

CONTACTS AND LOCATIONS:
Locations (1):
- Cankırı Karatekin University, Çankırı, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD often contains sensitive personal information about participants. Sharing this data may compromise their privacy and violate ethical guidelines or legal regulations